1 de 4

Informed Consent Form

Tittle: Effects of Traditional Concurrent Training and Concurrent Training

Composed by Strength Training and Dance Classes in Functional Performance,

Cognitive Function and Quality of Life of Older Adults: a Randomized

**Controlled Clinical Trial** 

Number: NCT05859243

Date: 16, May, 2023

Dear Sir,

You are being invited to participate, as a volunteer, in the research "Effects of

traditional concurrent training and concurrent training composed of strength training

combined with dance classes on functional performance, cognitive function and

quality of life in the elderly". If you grant permission to participate, please sign at the

end of the document. Your participation is not mandatory and you may withdraw your

consent at any time.

Responsible Researcher: Dr. Eduardo Lusa Cadore

Phone: 51 991193651

**Institution:** Federal University of Rio Grande do Sul - UFRGS

**Objectives:** To analyze the effects of traditional concurrent training and concurrent

training consisting of strength training combined with dance classes on functional

performance, cognitive function and quality of life in the elderly.

**Study procedures:** If you agree to participate in the research, you will be randomly

allocated to one of the following groups:

Traditional concurrent training group: Participants in this group will perform 30

minutes of weight training and 30 minutes of walking, twice a week over 12

weeks (three months). All training sessions will be held at ESEFID/UFRGS

with monitoring by qualified professionals.

Concurrent training group consisting of strength training combined with dance

classes: participants in this group will perform 30 minutes of weight training and 30 minutes of dance classes, twice a week over 12 weeks (three months). All training sessions will be held at ESEFID/UFRGS with monitoring by qualified professionals.

 Control group: participants in this group should maintain their usual routine for 12 weeks and, after this period, they will be able to choose to participate in one of the physical exercise groups according to their preference.

In addition, you will carry out the following evaluation procedures: (1) a questionnaire to assess the level of physical activity, (2) a questionnaire to assess mental health, (3) a sociodemographic characterization questionnaire, (4) a questionnaire to assess quality of life, (5) a test to assess cognitive performance, (6) a blood sample to assess the lipid profile, (7) a physical assessment, (8) eight physical tests to assess functional performance, and (9) a questionnaire to assess the affectivity of the intervention. All evaluations will be carried out by researchers from the School of Physical Education, Physiotherapy and Dance at UFRGS, except for the blood collection that will be carried out by a qualified researcher at the Laboratory of Memory Dysfunctions at UFRGS.

Risks and Discomforts: Research offers you more than minimal risk. The physical tests and training may cause some discomfort, fatigue or muscle damage, which will be avoided by familiarizing yourself with the exercises, warming up beforehand, offering rest and water, as well as monitoring by a qualified researcher. Blood collections may cause small skin lesions, however, it will be performed by a trained professional seeking to minimize this factor. All procedures may cause physical and mental fatigue due to the large number of questionnaires and evaluations performed. In this sense, to minimize this risk in all procedures, you will be asked periodically about your physical and mental state and, if you experience any symptoms of discomfort, a break will be held in an appropriate place. If there is any incident, the researcher in charge will be responsible for you and will accompany you in the care that is necessary. You will have the right to seek compensation for any damages resulting from the research.

Cost/reimbursement for the participant: We inform you that you will not incur any expenses arising from your participation and you will not receive any kind of gratuity

due to your participation in the research. Travel to the research sites can be carried out free of charge through the free pass system for seniors proposed by the City Hall of Porto Alegre - RS.

**Benefits:** You will have access to an individual report with the results of all the tests you perform during the study. These data can be used to support future physical training, in addition to serving as an indicator of health status. In addition, you will benefit from the physiological and functional adaptations provided by training.

**Other information:** The data used in this project will be used exclusively for the purposes of this study and all information will maintain the anonymity of the participants. Blood samples will be used only for this research and, at the end of the study, will be discarded. The data collected will be used only for the purposes of research and publication and will be kept for a period of 5 years before being destroyed.

Contact: At any time, you can request clarifying information about the study by e-mail: edcadore@yahoo.com.br, eduardarambo@gmail.com or by phone: 51 991193651 (Prof. Dr. Eduardo Lusa Cadore), 51 999079773 (Prof. Eduarda Blanco Rambo). Possible doubts regarding the ethical aspects of the research can be clarified directly at the Ethics and Research Committee – CEP of UFRGS, by e-mail: etica@propesq.ufrgs.br; by phone: (51) 3308-3787; or at the address Av. Paulo Gama, 110, Room 311, Annex I Building of the Rectory - Centro Campus, Porto Alegre/RS, from Monday to Friday, from 8:00 am to 12:00 pm and from 1:30 pm to 5:30 pm. The CEP is a collegiate body, with an advisory, deliberative and educational character, whose purpose is to evaluate, issue an opinion and monitor research projects involving human beings, in their ethical and methodological aspects, carried out within the scope of the institution.

| Participant Signature: | | |
|------------------------|---|---|
| Researcher: | | |
| Place and date: | / | 1 |